CLINICAL TRIAL: NCT01932203
Title: A Multicenter, Randomized, Double Blind Study to Compare the Efficacy Between Cilostazol and Aspirin on White Matter Changes by Cerebral Small Vessel Disease
Brief Title: Efficacy Study of Cilostazol and Aspirin on Cerebral Small Vessel Disease
Acronym: Challenge
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Inha University Hospital (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Principal Investigator, Inha University Hospital, Professor, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130006
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Small Vessel Disease
Keywords: Cerebral small vessel disease; Leukoaraiosis; Magnetic Resonance Imaging; Diffusion Tensor Imaging
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Leukoaraiosis | interventions — Aspirin; Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aspirin (Active Comparator): aspirin 100mg by mouth once a day for 104 weeks
  Interventions: Drug: aspirin
- Cilostazol (Experimental): Pletaal SR 200mg by mouth once a day for 104 weeks
  Interventions: Drug: cilostazol

INTERVENTIONS:
Drug: aspirin — 100mg once a day
  Arms: aspirin
Drug: cilostazol — 200mg once a day
  Other Names: Pletaal SR
  Arms: Cilostazol

SUMMARY:
There may be a difference in efficacy of cilostazol and aspirin on progression of white matter changes in cerebral small vessel disease.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the efficacy of aspirin and cilostazol on volume of white matter changes in cerebral small vessel disease.

The secondary objectives are to compare the impact of aspirin and cilostazol on DTI parameters, lacune, microbleeds, brain atrophy, cognition, depression, neurologic signs, gait, urination, and activities of daily living.

We also investigate risk factors associated with progression of cerebral small vessel disease.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 85 years of age
* He/She can walk to the hospital (walker or cane is permissible).
* Cerebral small vessel disease is observed on brain MRI.

  1) presence of one or more lacunar infarction and 2) moderate or severe confluent leukoaraiosis (defined as grade 2 or 3 on a modified Fazekas scale): periventricular WMCs with cap or rims lager than 5mm and deep subcortical WMCs >10 mm in maximum diameter
* written informed consent

Exclusion Criteria:

* Any patient with contraindication of antiplatelets
* Any patient with cardioembolic source
* Carotid bruit or large cerebral artery stenosis >50%
* Cortical infarction or subcortical infarction lager than 1.5 cm
* bleeding tendency
* chronic liver disease (AST or ALT >100 IL/L)
* chronic renal disease (Creatinine >3.0mg/dL)
* active gastrointestinal ulcer
* any patients with any severe or unstable medical disease that may prevent them from completing study requirements (i.e., unstable or severe asthma)
* Anemia (Hb <10g/dL) or thrombocytopenia
* Cardiac pacemaker or contraindication to MRI
* Pregnancy or breast-feeding
* drug or alcohol addiction
* Any other white matte disease (i.e., Multiple sclerosis, sarcoidosis, or brain irradiation, etc) or brain tumor
* Parkinson's disease, Alzheimer's disease or any other neurodegenerative disease
* any hearing or visual impairment that can disturb the efficient evaluation of the patient
* recent cerebral infarction with 3 months

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2013-07-17 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Volume of white matter changes (WMCs) | baseline, week 104
  Measure change of WMC on brain MRI

SECONDARY OUTCOMES:
Mean diffusivity (MD) and Fraction Anisotropy (FA) on Diffusion Tensor Imaging | baseline and week 104
  High MD and low FA means tissue damage.
Number of lacunes | baseline and week 104
  High number means tissue damage.
number of microbleeds | baseline and week 104
  High number means tissue damage.
brain volume and cortical thickness | baseline and week 104
  Low score means tissue damage.
Mini-Mental State Examination | baseline, week 52, and week 104
  Measure global cognition. Score range is 0-30. Higher score means good cognition.
Neurocognitive test | baseline, week 52, and week 104
  Seoul Verbal Learning Test, Boston Naming test-short form, ROCF copy, animal fluency, phonemic fluency, Stroop test, Digit-symbol test, Trail making test
Clinical Dementia Rating scale-sum of boxes | baseline, week 52, and week 104
  Measure global cognition. Score range is 0-18. Higher score means good cognition.
King's Health Questionnaire | baseline, week 42, and week 104
  Measure voiding function. Higher score means bad function.
Geriatric Depression Scale-Short form | baseline, week 52, and week 104
  Measure depression. Score range is 0-15. Higher score means depression.
Caregiver-Administered Neuropsychiatric Inventory (CGA-NPI) | baseline, week 52, and week 104
  Measure abnormal behavior. Score range is 0-144. Higher score means severe abnormal behavior.
Bayer Activities of Daily Living | baseline, week 52, and week 104
  Measure instrumental activities of daily living (ADL). Score range is 1-10. Higher score means bad ADL.
Barthel Index | baseline, week 52, and week 104
  Measure physical ADL. Score range is 0-20. Higher score means good physical ADL.
Pyramidal and Extrapyramidal Scale (PEPS) | baseline, week 52, and week 104
  Measure neurologic signs. Score range is 0-60. Higher score means many abnormal neurologic signs.
Timed UP and Go (TUG) test | basline, week 52, and week 104
  Measure gait. Higher score means bad gait.
Adverse event | baseline, week 4, 16, 28, 40, 52, 64, 76, 88, and 104
  measure any adverse events

OTHER OUTCOMES:
All ischemic stroke event | week 104
  cerebral infarction and transient ischemic attack
All vascular events | week 104
  including ischemic stroke, transient ischemic attack, myocardial infarction, angina pectoris, cerebral venous thrombosis, pulmonary embolism, symptomatic deep vein thrombosis, symptomatic peripheral artery occlusion, other vascular occlusion, and any revascularization procedure

CONTACTS AND LOCATIONS:
Overall Officials: Seong Hye Choi, MD, PhD, Principal Investigator — Inha University Hospital
Locations (19):
- South Korea (19):
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - National Health Insurance Corporation Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Dongtan Sacred Heart Hospital, Hallym University College of Medicine, Hwaseong-si, Gyeonggi-do
  - Wonkwang University Iksan Hospital, Iksan, Jeollabuk-do
  - Hallym University Medical Center, Anyang
  - Bucheon St.Mary's Hospital, Bucheon-si
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Eulji University School of Medicine, Daejeon
  - Konyang University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Gachon University Gil Medical, Incheon
  - Dong-A University Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Chungang University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Kwan J, Hafdi M, Chiang LLW, Myint PK, Wong LS, Quinn TJ. Antithrombotic therapy to prevent cognitive decline in people with small vessel disease on neuroimaging but without dementia. Cochrane Database Syst Rev. 2022 Jul 14;7(7):CD012269. doi: 10.1002/14651858.CD012269.pub2. PMID 35833913
- [Derived] Kim BC, Youn YC, Jeong JH, Han HJ, Kim JH, Lee JH, Park KH, Park KW, Kim EJ, Oh MS, Shim Y, Lee JM, Choi YH, Park G, Kim S, Park HY, Yoon B, Yoon SJ, Cho SJ, Park KC, Na DL, Park SA, Choi SH. Cilostazol Versus Aspirin on White Matter Changes in Cerebral Small Vessel Disease: A Randomized Controlled Trial. Stroke. 2022 Mar;53(3):698-709. doi: 10.1161/STROKEAHA.121.035766. Epub 2021 Nov 16. PMID 34781708
- [Derived] Han HJ, Kim BC, Youn YC, Jeong JH, Kim JH, Lee JH, Park KH, Park KW, Kim EJ, Oh MS, Shim YS, Park HY, Yoon B, Yoon SJ, Cho SJ, Park KC, Na DL, Park SA, Lee JM, Choi SH. A Comparison Study of Cilostazol and Aspirin on Changes in Volume of Cerebral Small Vessel Disease White Matter Changes: Protocol of a Multicenter, Randomized Controlled Trial. Dement Neurocogn Disord. 2019 Dec;18(4):138-148. doi: 10.12779/dnd.2019.18.4.138. Epub 2019 Dec 13. PMID 31942173